CLINICAL TRIAL: NCT04391777
Title: Determine the Effect of the Fourth Ventricle Compression Technique on Heart Rate, Respiratory Rate, Blood Pressure, Thermal Variation and Skin Conductivity in Healthy Young Adults: a Randomized Clinical Study
Brief Title: Determine the Effect of the Fourth Ventricle Compression Technique on Physiological Variables
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Natália Maria Oliveira Campelo, Professor, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OST1- 002
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Healthy Young Adults
Keywords: Osteopathy; Fourth ventricle compression technique; Physiological variables
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CV-4 group (Experimental): The initial selection will be made through a questionnaire, in order to fulfill the exclusion and inclusion criteria. On the data collection day a more detailed survey is performed and informed consent is signed.
  The patient waits for 5 minutes in the supine position, after which the baseline evaluation is performed.
  The CV-4 technique is performed following immediate evaluation. 15 minutes after the technique, a new evaluation of the variables is accomplished.
  Interventions: Other: Fourth ventricle compression technique (CV-4)
- Control group (Sham Comparator): The initial selection will be made through a questionnaire, in order to fulfill the exclusion and inclusion criteria. On the data collection day a more detailed survey is performed and informed consent is signed.
  The patient waits for 5 minutes in the supine position, after which the baseline evaluation is performed.
  The sham technique is performed following immediate evaluation. 15 minutes after the technique, a new evaluation of the variables is accomplished.
  Interventions: Other: Sham

INTERVENTIONS:
Other: Fourth ventricle compression technique (CV-4) — The participant is in the supine position and the principal investigator is seated at the patient's head, with elbows resting on the table. The main investigator overlaps his hands with the thenar eminences, contacting the occipital bone squamous part, between the external occipital protuberance and the participant's occipito-mastoid suture. The technique begins with a maintained compression on the occipital squamous part during a deep thorax exhalation. Throughout the compression of the occipital bone and the participant's voluntary inspirations, the principal investigator feels a gradual pressure increase at the thenar eminences. The technique will be performed until reaching the still point, in which the mobility of the occipital bone, respiratory rate and muscle tone decrease, or until 5 minutes elapsed.
  Arms: CV-4 group
Other: Sham — The main investigator uses the technique contact but does not perform any type of tissue traction or compression, maintaining this contact for 5 minutes. At the end of the stipulated time, the contact is removed in a subtle way.
  Arms: Control group

SUMMARY:
This study aims to analyze the influence of the fourth ventricle compression technique in heart rate, respiratory rate, blood pressure, conductivity and thermal variability of the skin in healthy young adults.

DETAILED DESCRIPTION:
The fourth ventricle compression technique (CV-4) is one of the most important techniques in the treatment of cranial osteopathy.

During the present study, the effects of CV-4 technique will be analyzed in the following variables: heart rate, respiratory rate, blood pressure, conductivity and thermal variation of the skin.

According to the literature, CV-4 technique will cause changes in all of the studied variables, except the respiratory rate, through the activation of the brain stem, namely the parasympathetic nerve centers.

Regarding the respiratory rate, it is justified by the fourth ventricle and the respiratory centers proximity.

Concerning heart rate and respiratory rate, during the CV-4 technique the literature describes a decrease in the values of this variables. However, other studies refer that the technique does not produce relevant effects in the heart and respiratory rates variation, probably because there was no stipulated time to finish the technique, ending subjectively compared to previous ones.

When it comes to blood pressure, a decrease in systolic blood pressure values is noticed by some authors.

In which concerns the variation in body temperature, according to the literature, there were no significant results obtained when performing CV-4.

During the performed literature analysis,there were not found any studies concerning the influences of the CV-4 technique in the thermal conductivity variable.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants aged between 18 and 33 years.

Exclusion Criteria:

* Cognitive deficits that can possibly compromise the understanding of the study instructions;
* Any type of medication taken that may have influences at the variables under study in the previous 7 days;
* Cranio-cervical injuries, surgery to the skull and /or spine in the last 12 months;
* Chronic cardiorespiratory, renal, systemic, neurological, musculoskeletal, oncological and psychiatric pathologies;
* Headaches, migraines, dizziness and / or nausea while performing the techniques;
* Caffeine and / or alcohol intake in the 6 hours prior to the data collection;
* Tobacco consumption in the 30 minutes prior to the data collection;
* Practice of intense physical exercise in the 90 minutes prior to the data collection;
* Pregnant women or menstruating;
* Participants who were submitted to manual therapy treatments during the past month;
* Osteopathy students of 3rd year or higher degree, in order to prevent the participant from recognizing which group they belong to.

Ages: 18 Years to 33 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in heart rate variability immediately after the intervention | Immediately after the intervention.
  To obtain the heart rate measurements, a pulse volume sensor (Biosignalsplux researcher) was connected to the third finger of the hand, with the patient lying supine. The sensor was only removed after completing all the evaluation moments.
Change from Baseline in heart rate variability 15 minutes after the intervention | 15 minutes after the intervention.
  To obtain the heart rate measurements, a pulse volume sensor (Biosignalsplux researcher) was connected to the third finger of the hand, with the patient lying supine. The sensor was only removed after completing all the evaluation moments.

SECONDARY OUTCOMES:
Change from Baseline in respiratory rate variability immediately after the intervention | Immediately after the intervention.
  To obtain the respiratory rate measurements, a respiratory belt transducer (Biopac Systems) was adjusted to the patient's thorax, at the xiphoid process level, with the patient lying supine. The sensor was only removed after completing all the evaluation moments.
Change from Baseline in respiratory rate variability 15 minutes after the intervention | 15 minutes after the intervention
  To obtain the respiratory rate measurements, a respiratory belt transducer (Biopac Systems) was adjusted to the patient's thorax, at the xiphoid process level, with the patient lying supine. The sensor was only removed after completing all the evaluation moments.
Change from Baseline in blood pressure variability immediately after the intervention | Immediately after the intervention.
  To obtain the blood pressure measurements, a digital sphygmomanometer was applied to the patient's left arm, with the patient lying supine. The sensor was only removed after completing all the evaluation moments.
Change from Baseline in blood pressure variability 15 minutes after the intervention | 15 minutes after the intervention.
  To obtain the blood pressure measurements, a digital sphygmomanometer was applied to the patient's left arm, with the patient lying supine. The sensor was only removed after completing all the evaluation moments.
Change from Baseline in skin conductivity variability immediately after the intervention | Immediately after the intervention.
  To obtain the skin conductivity measurements, 2 electrodermal activity sensors (Biosignalsplux researcher) were connected to the patient's first finger, on the carpometacarpal and metacarpophalangeal joints, with the patient lying supine. The sensor was only removed after completing all the evaluation moments.
Change from Baseline in skin conductivity variability 15 minutes after the intervention | 15 minutes after the intervention.
  To obtain the skin conductivity measurements, 2 electrodermal activity sensors (Biosignalsplux researcher) were connected to the patient's first finger, on the carpometacarpal and metacarpophalangeal joints, with the patient lying supine. The sensor was only removed after completing all the evaluation moments.
Change from Baseline in skin thermal variation immediately after the intervention | Immediately after the intervention.
  To obtain the skin thermal variation measurements, negative temperature coefficient (NTC) thermistor sensors (Biosignalsplux researcher) were connected to the patient's first finger, on the carpometacarpal and metacarpophalangeal joints, with the patient lying supine. The sensor was only removed after completing all the evaluation moments.
Change from Baseline in skin thermal variation 15 minutes after the intervention | 15 minutes after the intervention.
  To obtain the skin thermal variation measurements, negative temperature coefficient (NTC) thermistor sensors (Biosignalsplux researcher) were connected to the patient's first finger, on the carpometacarpal and metacarpophalangeal joints, with the patient lying supine. The sensor was only removed after completing all the evaluation moments.

CONTACTS AND LOCATIONS:
Overall Officials: Natália MO Campelo, Principal Investigator — Escola Superior de Saúde do Politécnico do Porto
Locations (1):
- Escola Superior da Saúde do Porto, Porto, Portugal

REFERENCES:
- [Result] Jakel A, von Hauenschild P. Therapeutic effects of cranial osteopathic manipulative medicine: a systematic review. J Am Osteopath Assoc. 2011 Dec;111(12):685-93. PMID 22182954
- [Result] Cardoso-de-Mello-E-Mello-Ribeiro AP, Rodriguez-Blanco C, Riquelme-Agullo I, Heredia-Rizo AM, Ricard F, Oliva-Pascual-Vaca A. Effects of the Fourth Ventricle Compression in the Regulation of the Autonomic Nervous System: A Randomized Control Trial. Evid Based Complement Alternat Med. 2015;2015:148285. doi: 10.1155/2015/148285. Epub 2015 Jun 14. PMID 26199632
- [Result] Milnes, K., & Moran, R. W. (2007). Physiological effects of a CV4 cranial osteopathic technique on autonomic nervous system function: A preliminary investigation. International Journal of Osteopathic Medicine, 10(1), 8-17. https://doi.org/10.1016/j.ijosm.2007.01.003
- [Result] Cutler MJ, Holland BS, Stupski BA, Gamber RG, Smith ML. Cranial manipulation can alter sleep latency and sympathetic nerve activity in humans: a pilot study. J Altern Complement Med. 2005 Feb;11(1):103-8. doi: 10.1089/acm.2005.11.103. PMID 15750368
- [Result] Miana L, Bastos VH, Machado S, Arias-Carrion O, Nardi AE, Almeida L, Ribeiro P, Machado D, King H, Silva JG. Changes in alpha band activity associated with application of the compression of fourth ventricular (CV-4) osteopathic procedure: a qEEG pilot study. J Bodyw Mov Ther. 2013 Jul;17(3):291-6. doi: 10.1016/j.jbmt.2012.10.002. Epub 2012 Nov 16. PMID 23768271
- [Result] Curi ACC, Maior Alves AS, Silva JG. Cardiac autonomic response after cranial technique of the fourth ventricle (cv4) compression in systemic hypertensive subjects. J Bodyw Mov Ther. 2018 Jul;22(3):666-672. doi: 10.1016/j.jbmt.2017.11.013. Epub 2017 Dec 9. PMID 30100295
- [Result] Bayo-Tallon V, Esquirol-Caussa J, Pamias-Massana M, Planells-Keller K, Palao-Vidal DJ. Effects of manual cranial therapy on heart rate variability in children without associated disorders: Translation to clinical practice. Complement Ther Clin Pract. 2019 Aug;36:125-141. doi: 10.1016/j.ctcp.2019.06.008. Epub 2019 Jul 2. PMID 31383430